CLINICAL TRIAL: NCT04691401
Title: Impact of AI (Artificial Intelligence) on Adenoma Detection During Colonoscopy in FIT+ Patients: a Prospective Randomized Controlled Trial
Brief Title: Impact of Artificial Intelligence (AI) on Adenoma Detection During Colonoscopy in FIT+ Patients.
Acronym: AIFIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Valduce Hospital (Other)
Responsible Party: Principal Investigator, Franco Radaelli, Head of Gastroenterology Unit, Valduce Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 598/2020
Record Dates: First submitted 2020-12-17; First posted 2020-12-31 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Polyp of Colon
Keywords: adenoma detection
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard WL (white light) colonoscopy (No Intervention): all patients receive standard colonoscopy (with high definition- HD- endoscopes) with white light (WL) in both insertion and withdrawal phase; all polyps identified are removed and sent for histopathology examination.
- Standard colonoscopy with assistance of Artificial Intelligence (CAD-EYE (Fujifilm Co, Tokyo, Japan) (Experimental): all patients receive colonoscopy examinations (with HD endoscopes) equipped with an Ai system (CAD-EYE, Fujifilm Co, Tokyo, Japan) in both insertion and withdrawal phase). This system is a real-time computer-assisted image analysis that allows automatic polyp identification without modifications to the colonoscope or to the actual endoscopic procedure. When CAD EYE identifies a polyp, both a visual (a green blinking box surrounding the identified polyp, called the detection box) and an acoustic alarm pop up and attract the endoscopist attention. Around the endoscopic image a visual assist circle is shown and lights up in the direction where the suspicious polyp is detected.All polyps identified are removed and sent for histopathology examination.
  Interventions: Device: Artificial Intelligence System (CAD EYE, Fujifilm Co.)

INTERVENTIONS:
Device: Artificial Intelligence System (CAD EYE, Fujifilm Co.) — A dedicated CNN-based AI system (CAD EYE, Fujifilm Co, Tokyo, Japan) has been recently developed. The Computer-aided diagnosis (CAD) CAD EYE system is a real-time computer-assisted image analysis that allows automatic polyp identification without modifications to the colonoscope or to the actual endoscopic procedure. When CAD EYE identifies a polyp, both a visual (a green blinking box surrounding the identified polyp, called the detection box) and an acoustic alarm pop up and attract the endoscopist attention. Around the endoscopic image a visual assist circle is shown and lights up in the direction where the suspicious polyp is detected.
  Arms: Standard colonoscopy with assistance of Artificial Intelligence (CAD-EYE (Fujifilm Co, Tokyo, Japan)

SUMMARY:
The Italian screening program invites the resident population aged 50-74 for Fecal Immunochemical Test (FIT) every 2 years. Subjects who test positive are referred for colonoscopy. Maximizing adenoma detection during colonoscopy is of paramount importance in the framework of an organized screening program, in which colonoscopy represent the key examination. Initial studies consistently show that Artificial iIntelligence-based systems support the endoscopist in evaluating colonoscopy images potentially increasing the identification of colonic polyps. However, the studies on AI and polyp detection performed so far are mostly focused on technical issues, are based on still images analysis or recorded video segments and includes patients with different indications for colonoscopy. At the best of our knowledge, data on the impact on AI system in adenoma detection in a FIT-based screening program are lacking. The present prospective randomized controlled trial is aimed at evaluating whether the use of an AI system increases the ADR (per patient analysis) and/or the mean number of adenomas per colonoscopy in FIT-positive subjects undergoing screening colonoscopy. Therefore Patients fulfilling the inclusion criteria are randomized (1:1) in two arms: A) patients receive standard colonoscopy (with high definition-HD endoscopes) with white light (WL) in both insertion and withdrawal phase; all polyps identified are removed and sent for histopathology examination; B) patients receive colonoscopy examinations (with HD endoscopes) equipped with an AI system (in both insertion and withdrawal phase); all polyps identified are removed and sent for histopathology examination. In the present study histopathology represents the reference standard.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive adult (50-74 yrs.) outpatients undergoing colonoscopy in the frame of the FIT-based screening program.

Exclusion Criteria:

* patients with CRC history or hereditary polyposis syndromes or hereditary non-polyposis colorectal cancer
* patients with inadequate bowel preparation
* patients in which cecal intubation was not achieved or scheduled for partial examinations
* patients with gastrointestinal symptoms
* polyps could not be resected due to ongoing anticoagulation preventing resection and pathological assessment

Ages: 50 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Actual)
Dates: Start 2020-12-20 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
ADR | 10 months
  Adenoma Detection Rate: rate of participants with at least on adenoma detected during colonoscopy
APC | 10 months
  Adenoma per Colonoscopy: it is determined by dividing the total number of adenomas removed by the total number of colonoscopies performed

SECONDARY OUTCOMES:
Adv-ADR | 10 months
  Adv-ADR: rate of participants with at least on advanced adenoma detected during colonoscopy
SSL-DR: | 10 months
  SSL-ADR: the serrated lesions with neoplastic potential (sessile serrated lesions-SSA; traditional serrated adenomas - TSA) detection rate.

OTHER OUTCOMES:
Impact of Ai on endoscopist with different ADR | 10 months
  The variation in ADR will be stratified according the initial ADR of endoscopists participating in the present study

CONTACTS AND LOCATIONS:
Locations (1):
- Gastroenterology Unit, Valduce Hospital, Como, Italy

IPD SHARING:
Plan to Share IPD: No